CLINICAL TRIAL: NCT06941233
Title: Our Peers - Empowerment and Navigational Support - Community Living (OP-ENS - CL)
Brief Title: Our Peers - Empowerment and Navigational Support - Community Living: Remote Peer Navigator Intervention for Adults With Newly Acquired Disabilities Transitioning to Community Living (OP-ENS -CL)
Acronym: OP-ENS - CL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Susan Magasi (Other)
Collaborators: Northwestern University Feinberg School of Medicine (Other); Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor-Investigator, Susan Magasi, Professor, University of Illinois at Chicago
Organization: University of Illinois at Chicago (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2025-0397; 90RTCP0005-01-00 (Other Grant/Funding Number: National Institute on Disability, Independent Living and Rehabilitation Research)
Record Dates: First submitted 2025-04-15; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Disabled Persons
Keywords: peer navigators; community health worker

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention or usual care groups using block randomization with randomly selected blocks of 4, 8, or 12. Randomization sequence will be generated using SAS algorithm.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the nature of the intervention it is not possible to mask participants and interventionists to group assignment. Outcome assessor and investigators will be unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OP-ENS - CL Intervention (Experimental): Participants will be matched with a peer navigator. As part of this complex behavioral intervention, participants and peer navigators will engage in a systematic process of barrier and strength identification, goal setting and action planning related to issues of healthcare access and quality. Participants and peers will meet remotely at least monthly over the course of the 12-month study period (but frequency is determined by participant need). Given the nature of the disability and community living experience, we anticipate the needs and therefore frequency will fluctuate over the duration of the study period. Beginning in month 10, participants and peers will engage in a period of transition planning to ensure that participants have the strategies and supports in place to assume the role of their own navigator.
  Interventions: Behavioral: Our Peers - Empowerment and Navigational Support - Community Living (OP-ENS - CL)
- Usual Care (No Intervention): Participants randomized to the usual care group will continue with their usual health, healthcare, and community living services routines. Participants in the usual care group will receive a monthly newsletter with general interest information relevant to the disability community.

INTERVENTIONS:
Behavioral: Our Peers - Empowerment and Navigational Support - Community Living (OP-ENS - CL) — Op-ENS - CL is a 12-month, remote delivered peer navigator intervention. Participants will meet with a trained peer navigator who mentors nad supports them through a manualized process of collaborative conversations, barrier identification, asset mapping, goal setting, and action planning along with on-going social support and information sharing.
  Arms: OP-ENS - CL Intervention

SUMMARY:
The goal of this clinical trial is to learn if a remote peer navigator intervention (OP-ENS - CL) for people with newly acquired physical disabilities returning to community living after rehabilitation improves self-reported social support, health, and community participation. The main questions it aims to answer are:

Do people with acquired physical disabilities who receive the remote peer navigator intervention experience greater social support and self-efficacy than people in the control group?

Do people with acquired physical disabilities who receive the remote peer navigator intervention have better self-reported health and social participation outcomes than people in the control group?

Is the OP-ENS - CL intervention acceptable to people with newly acquired physical disabilities returning to community living?

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy and social validity of the OP-ENS - CL (Our Peers - Empowerment and Navigational Support - Community Living) a remote 12-month peer navigator intervention using a clinical trial design in a sample of adults with newly acquired with physical disabilities transitioning to community living.

Participants will be recruited through community and clinical networks and screened for eligibility. Participants will be randomly assigned to either the intervention or usual care groups. Participants in the intervention group will be matched with a trained peer health navigator (who is also a person with a physical disability). Using a structure process of barrier identification, goal setting and action planning peer health navigators will work with participants to help address their healthcare needs and concerns, including such things as patient-provider communication, transportation, access to durable medical equipment. It is important to note that peer health navigators are not healthcare providers and do not provide medical or health advice. Participants in the intervention trial are asked to meet with their peer navigator at least once a month during the study period. To encourage participation in this intervention, progressive micro-incentives are integrated into the study protocol. To promote equipoise, a similar micro-incentive schedule is created for the usual care group.

Data Collection - All participants, regardless of group assignment, will be interviewed at 3 time points (baseline, 6 months, 13 months) using a self-report measures of healthcare access, quality, and outcomes as well as measures of social support and patient activation. Data collectors will be blinded to group assignment and not involved in the delivery of the OP-ENS - CL intervention.

Data Analysis - The investigators will employ mixed effects model using each study outcome as a time-varying dependent variable and treatment group (PHN vs. usual care) as the main fixed effect. Baseline characteristics including race/ethnicity, gender, and socioeconomic status will be entered as time-invariant covariates if baseline group differences are observed (in spite of randomization). Subject intercept will be modeled as a random effect. The null hypothesis will be rejected if a significant group*time interaction effect is observed. The investigators hypothesize that PN will have a more favorable trajectory slope of study outcomes than the matched control group. For each hypothesis, post-hoc analysis will be conducted to assess difference in each outcome variable between the two groups at different time points. The mixed models will run using PROC MIXED from of SAS 9.3 (Cary, NC). The method of estimation will be maximum likelihood (ML). A variety of covariance structures (first order regressive, compound symmetry, toeplitz, variance components, unstructured) will be carefully examined and compared for best model fit, Akaike's Information (AIC) and Bayesian Information Criteria (BIC). These statistics are functions of the log likelihood and can be compared across models. As missing data are inevitable in a longitudinal study, values will be imputed where possible using either mean (median) substitute or formal imputation procedures such as EM algorithm if missing data are MCAR (missing completely at random) or MAR (missing at random). If missing data are NMAR (not missing at random), the "pattern mixture" approach will be used to compute a "weighted average" of the parameters that are associated with the missing data to estimate what the data would have been.

ELIGIBILITY:
Inclusion Criteria: 1) Self-identify as a person with physical disability due to a neurological condition, including SCI, stroke, TBI, multiple sclerosis, or Parkinson's disease (according to the American Community Survey 6-Items), 2) onset of disability within the last 6 months, 3) transitioned to community living in the past 4 months, 4) able to speak, read and understand English, 5) own or have regular access to either a smartphone (Android or iOS operating system), tablet, laptop, or desktop computer with internet access. 6) adults 18 years of age or older, 7) able to provide informed consent.

Exclusion Criteria: 1) Cognitive, sensory, or physical functional limitations that interfere with effective use of the OP-ENS - CL app.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure | Baseline, 6 months, 13 months.
  The 13-item self-report measure assesses perceived knowledge, skills, and confidence for self-management
PROMIS Self-Efficacy Short Form | Baseline, 6 months, 13 months.
  4-item self-report short form measure assessing confidence in one's ability to perform specific tasks or behaviors
PROMIS Emotional Support, short form | Baseline, 6 months, 13 months.
  8-item self-report short forms assessing the availability of 3 types of emotional support
PROMIS informational support, short form | Baseline, 6 months, 13 months.
  8-item self-report short forms assessing the availability of informational support
PROMIS Instrumental Support, short form | Baseline, 6 months, 13 months.
  8-item self-report short forms assessing the availability of instrumental support

SECONDARY OUTCOMES:
PROMIS Global Health | Baseline, 6 months, 13 months.
  8-item self-report short form assessing perceived physical, mental, and social health.
PROMIS Depression | Baseline, 6 months, 13 months.
  8-item short form assessing self-reported affect, views of self, social cognition, and decreased positive affect
PROMIS Ability to Participate in Social Roles and Activities | Baseline, 6 months, 13 months.
  8-item short form assessing perceived ability to perform one's usual social roles and activities
Community Participation Indicators, Enfranchisement Scale | Baseline, 6 months, 13 months.
  19-item self-report measures 3 subjective domains of participation, choice and control, contributing to one's community, and feeling valued.
Canadian Occupational Performance Measure | Baseline, 6 months, 13 months.
  Semi-structured interview including 5 step process to identify subjects' goals. Subjects rate their perceived performance and satisfaction on 1 - 5 goals.

OTHER OUTCOMES:
Patient Satisfaction with Logistical Aspects of Navigation Scale | 13-month
  Forty eight item self-report measure of patient's satisfaction with a medical navigator's help with logistical issues related to care.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Magasi, PhD, Principal Investigator — University of Illinois Chicago
Locations (1):
- University of Illinois Chicago, Department of Occupational Therapy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
To preserve the privacy and confidentiality of study participants, we may elect not to share the IPD.

REFERENCES:
- [Background] Magasi S, Papadimitriou C, Panko Reis J, The K, Thomas J, VanPuymbrouck L, Wilson T. Our Peers-Empowerment and Navigational Support (OP-ENS): Development of a Peer Health Navigator Intervention to Support Medicaid Beneficiaries With Physical Disabilities. Rehabil Process Outcome. 2019 Apr 26;8:1179572719844759. doi: 10.1177/1179572719844759. eCollection 2019. PMID 34497460
- [Background] Magasi S, Angell AM, Papadimitriou C, Ramirez RD, Ferlin A, Reis JP, Wilson T. Inside an Occupational Therapy-Disability Community Partnership to Promote Health Management: Ethnography of a Research Collaboration. Am J Occup Ther. 2021 Jul 1;75(4):7504180050p1-7504180050p12. doi: 10.5014/ajot.2021.045468. PMID 34780614
- See also: The Program for Healthcare Justice for People with Disabilities is the principal investigator, Susan Magasi, lab website. — https://hjpwd.ahs.uic.edu/
- Available data/document: Study Protocol — https://hjpwd.ahs.uic.edu — study protocol may be accessed by contacting the research team